CLINICAL TRIAL: NCT05296629
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Active and Placebo Controlled Study to Assess the Safety, Efficacy and Tolerability of Oral DFD-29 Extended Release Capsules for the Treatment of Inflammatory Lesions of Rosacea Over 16 Weeks.
Brief Title: A Randomized, Double-Blind Study to Assess the Safety, Efficacy and Tolerability of Oral DFD-29 Capsules for the Treatment of Rosacea.
Acronym: MVOR-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Journey Medical Corporation (Industry)
Collaborators: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DFD-29-CD-004
Record Dates: First submitted 2022-03-17; First posted 2022-03-25 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: A multicenter, randomized, parallel-group, double-blind, controlled study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DFD-29 (Experimental): DFD-29 (40 mg) extended release capsules
  Interventions: Drug: DFD-29
- Doxycycline 40 mg (Active Comparator): Doxycycline 40 mg modified release capsules
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Placebo capsules matching DFD-29
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DFD-29 — DFD-29 (40 mg) extended release capsules
  Arms: DFD-29
Drug: Doxycycline — Doxycycline 40 mg capsules
  Arms: Doxycycline 40 mg
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
This is a 16-week, multicenter, randomized, parallel-group, double-blind, controlled study. After assessing eligibility during a screening period of up to 30 days, approximately 320 subjects at least 18 years old who are diagnosed with moderate to severe papulopustular rosacea will be randomized in a 3:3:2 ratio to DFD-29 (40 mg), Doxycycline capsules 40 mg, or Placebo once daily for 16 weeks.

DETAILED DESCRIPTION:
This is a 16-week, multicenter, randomized, parallel-group, double-blind, controlled study. After assessing eligibility during a screening period of up to 30 days, approximately 320 subjects at least 18 years old who are diagnosed with moderate to severe papulopustular rosacea will be randomized in a 3:3:2 ratio to DFD-29 (40 mg), Doxycycline capsules 40 mg, or Placebo once daily for 16 weeks.

Subject visits are scheduled at Screening, Baseline (Day 1), and Weeks 2, 4, 8, 12, and 16. Clinical assessments of efficacy will be conducted based on Investigator's Global Assessment modified scale without erythema (IGA), Clinician's Erythema Assessment (CEA), and total inflammatory lesion count at Weeks 2, 4, 8, 12, and 16 compared to Baseline.

Laboratory assessments of blood (hematology and biochemistry) and urine (routine tests) will be conducted at Screening and Week 16 (end of study [EOS] or early termination) to assess for any changes in the safety parameters. Other safety assessments include vital signs, physical examination, urine pregnancy tests (for females of childbearing potential), and collection of AE data.

The impact of the treatment on the quality of life (QoL) of the subjects will be assessed using the rosacea-specific tool RosaQoL in addition to the Dermatology Life Quality Index (DLQI) at Baseline and Weeks 2, 4, 8, 12, and 16.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female subjects aged 18 years and above.
* Subjects must be in good general health as determined by the investigator and supported by the medical history.
* Subjects must have a clinical diagnosis of papulopustular rosacea with IGA grade 3 (moderate) or IGA grade 4 (severe) at Baseline.
* Subjects must have 15 to 60 (both inclusive) inflammatory lesions (papules and pustules) of rosacea over the face at Baseline.
* Subjects must have not more than 2 nodules or cysts at Baseline.

Key Exclusion Criteria:

* Female subjects who are pregnant or nursing or planning to become pregnant during the study.
* Male subjects whose female partner is planning to conceive a child.
* Clinically significant abnormal laboratory test results that, in the opinion of the investigator, would compromise the subject's safety or ability to participate in the trial.
* History of organ transplant requiring immunosuppression, HIV, or other immune compromised state.
* History of lupus-like syndrome, autoimmune hepatitis, vasculitis, or serum sickness.
* Any clinically significant condition or situation other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R Sidgiddi, M.D., Study Director — Journey Medical Corporation
Locations (27):
- United States (27):
  - Clinical Trial Site 05, Rogers, Arkansas
  - Clinical Trial Site 10, Cerritos, California
  - Clinical Trial Site 03, Fremont, California
  - Clinical Trial Site 25, San Diego, California
  - Clinical Trial Site 29, San Diego, California
  - Clinical Trial Site 11, Clearwater, Florida
  - Clinical Trial Site 08, Coral Gables, Florida
  - Clinical Trial Site 22, Coral Gables, Florida
  - Clinical Trial Site 02, Indianapolis, Indiana
  - Clinical Trial Site 27, Overland Park, Kansas
  - Clinical Trial Site 09, Brighton, Massachusetts
  - Clinical Trial Site 18, Ann Arbor, Michigan
  - Clinical Trial Site 28, Warren, Michigan
  - Clinical Trial Site 21, New Brighton, Minnesota
  - Clinical Trial Site 15, Las Vegas, Nevada
  - Clinical Trial Site 24, New York, New York
  - Clinical Trial Site 17, High Point, North Carolina
  - Clinical Trial Site 04, Wilmington, North Carolina
  - Clinical Trial Site 06, Beachwood, Ohio
  - Clinical Trial Site 01, Sugarloaf, Pennsylvania
  - Clinical Trial Site 19, East Greenwich, Rhode Island
  - Clinical Trial Site 23, Nashville, Tennessee
  - Clinical Trial Site 20, College Station, Texas
  - Clinical Trial Site 13, Houston, Texas
  - Clinical Trial Site 07, Plano, Texas
  - Clinical Trial Site 26, San Antonio, Texas
  - Clinical Trial Site 12, San Antonio, Texas

REFERENCES:
- [Derived] Bhatia N, Del Rosso J, Stein Gold L, Lain E, Draelos ZD, Sidgiddi S; MVOR-1 and MVOR-2 Study Investigators. Efficacy, Safety, and Tolerability of Oral DFD-29, a Low-Dose Formulation of Minocycline, in Rosacea: Two Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2025 May 1;161(5):499-507. doi: 10.1001/jamadermatol.2024.6542. PMID 40042869

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline 40 mg Capsule: Doxycycline 40 mg capsule administered once daily for 16 weeks
Period: Overall Study
Arm/Group | DFD-29 | Doxycycline 40 mg Capsule | Placebo
Started | 122 | 121 | 80
Completed | 117 | 98 | 73
Not Completed | 5 | 23 | 7
Not completed — Withdrawal by Subject | 3 | 10 | 4
Not completed — Lost to Follow-up | 2 | 7 | 1
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Protocol Violation | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: ITT Subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | DFD-29 | Doxycycline 40 mg Capsule | Placebo | Total
Number analyzed (Participants) | 122 | 121 | 80 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (13.16) | 46.7 (14.11) | 47.2 (14.09) | 47.2 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 90 | 63 | 247
  Male | 28 | 31 | 17 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 6 | 5 | 6 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 113 | 111 | 71 | 295
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 122 | 121 | 80 | 323
Investigators Global Assessment (IGA) grade [Count of Participants; unit: Participants] — The modified IGA scale is a 5-point scale from Grade 0 to Grade 4, wherein Grade 0 is Clear, Grade 1 is Near Clear, Grade 2 is Mild, Grade 3 is Moderate and Grade 4 is Severe Rosacea. A lowering of the score with treatment indicates an improvement in the disease condition and a beneficial outcome.
  Participants
    Moderate | 101 | 110 | 68 | 279
    Severe | 21 | 11 | 12 | 44
Total Inflammatory Lesion Count [Mean (Standard Deviation); unit: Lesion count] | 26.4 (10.46) | 23.8 (8.75) | 25.9 (8.84) | 25.3 (9.50)
Clinician's Erythema Assessment (CEA) score [Count of Participants; unit: Participants]
  0 = None | 0 | 0 | 0 | 0
  1 = Mild | 3 | 2 | 2 | 7
  2 = Moderate | 50 | 45 | 32 | 127
  3 = Significant | 57 | 61 | 37 | 155
  4 = Severe | 12 | 13 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA) Treatment Success Compared to Placebo.
Description: Proportion of subjects with IGA (modified scale without erythema) 'treatment success' - Grade 0 or 1 at Week 16 with at least 2 grade reduction from Baseline to Week 16, in the DFD-29 group compared to Placebo.
  The modified IGA scale is a 5-point scale from Grade 0 to Grade 4, wherein Grade 0 is Clear, Grade 1 is Near Clear, Grade 2 is Mild, Grade 3 is Moderate and Grade 4 is Severe Rosacea. A lowering of the score with treatment indicates an improvement in the disease condition and a beneficial outcome.
Time Frame: Baseline to Week 16.
Population: ITT population defined as, 'All randomized subjects'
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-29 | Placebo
Number analyzed (Participants) | 122 | 80
Participants | 79 | 25

2. Primary Outcome: Change in Total Inflammatory Lesion Count Compared to Placebo.
Description: Total inflammatory lesion count (sum of papules, pustules, and nodules) change from Baseline to Week 16, in the DFD-29 group compared to Placebo.
Time Frame: Baseline to Week 16.
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: lesions
Arm/Group | DFD-29 | Placebo
Number analyzed (Participants) | 122 | 80
lesions | -20.6 (0.77) | -11.4 (0.97)

3. Secondary Outcome: IGA Treatment Success Compared to Doxycycline.
Description: Proportion of subjects with IGA treatment success at week 16 in the DFD-29 group compared to Doxycycline capsules 40 mg.
Time Frame: Baseline to Week 16.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-29 | Doxycycline 40 mg
Number analyzed (Participants) | 122 | 121
Participants | 79 | 56

4. Secondary Outcome: Change in Total Inflammatory Lesion Count Compared to Doxycycline.
Description: Total inflammatory lesion count change from Baseline to week 16 in the DFD-29 group compared to Doxycycline capsules 40 mg.
Time Frame: Baseline to Week 16.
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: lesions
Arm/Group | DFD-29 | Doxycycline 40 mg
Number analyzed (Participants) | 122 | 121
lesions | -20.6 (0.69) | -15.6 (0.73)

5. Secondary Outcome: Clinician's Erythema Assessment (CEA) Compared to Placebo.
Description: Proportion of subjects with at least 2-grade reduction in CEA score from Baseline to Week 16 in the DFD-29 group compared to Placebo.
Time Frame: Baseline to Week 16.
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | DFD-29 | Placebo
Number analyzed (Participants) | 122 | 80
Participants | 39 | 11

ADVERSE EVENTS:
Time Frame: From the signing of informed consent up to 16 weeks of study treatment.
Description: AEs were collected by spontaneous reports from subjects, either verbal or recorded in the subject's diary, by directed questioning of subjects, and by observation.
  The number of participants at risk for safety assessments were drawn from the safety population. Hence, they are slightly different from the efficacy assessments where the ITT population was used.
Arm/Group | DFD-29 | Doxycycline 40 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/121 | 0/116 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/121 | 0/116 | 0/76
Other Adverse Events (participants affected / at risk) | 17/121 | 19/116 | 18/76
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFD-29 (N=121) | Doxycycline 40 mg (N=116) | Placebo (N=76)
COVID-19 (Infections and infestations) | 4 | 3 | 4
Nasopharyngitis (Infections and infestations) | 4 | 2 | 3
Vulvovaginal mycotic infections (Infections and infestations) | 2 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 0 | 4 | 2
Headache (Nervous system disorders) | 3 | 2 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 2 | 1
Gout (Metabolism and nutrition disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-06-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT05296629/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT05296629/SAP_001.pdf